CLINICAL TRIAL: NCT05834439
Title: The Effect of Flower Printing Activity Applied to the Elderly in the Nursing Home on the Anxiety Levels of the Elderly: A Single-Blind Randomized Controlled Study
Brief Title: Flower Print Activity Applied to the Elderly in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Assoc. Prof., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1Ordu
Record Dates: First submitted 2022-12-12; First posted 2023-04-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Elderly; Gardening; Anxiety; Nursing Caries
Keywords: Gardening, Floral print, Elderly, Anxiety, Nursing
MeSH Terms: conditions — Anxiety Disorders | interventions — Nursing Homes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group
  Interventions: Other: flower printing activities for the elderly
- Control group (Other): Control group
  Interventions: Other: Routine activities in nursing home

INTERVENTIONS:
Other: flower printing activities for the elderly — Experimental group
  Arms: Experimental group
Other: Routine activities in nursing home — Control group
  Arms: Control group

SUMMARY:
This research will be carried out in order to determine the effect of the flower pressure activity applied to the elderly in the nursing home on the anxiety levels of the elderly.

DETAILED DESCRIPTION:
This research will be carried out in order to determine the effect of the flower pressure activity applied to the elderly in the nursing home on the anxiety levels of the elderly.

Hypotheses H0 = Flower pressure activity applied to the elderly in the nursing home does not affect the anxiety level of the elderly.

H1= Flower pressure activity applied to the elderly in the nursing home reduces the anxiety level of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Has no physical handicap that may hinder the activity of flower printing,
* No vision or hearing loss that may hinder the activity of flower printing,
* Open to communication and cooperation,
* The elderly who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Have a serious medical disability,
* Having a serious psychiatric diagnosis,
* Severely demented and
* The elderly who do not want to continue the research will be excluded from the research.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Geriatric Anxiety Scale | day 0 and day 30
  The scale developed by Pachana et al. (2007) was adapted to Turkish by Pamir Akın (2010). The Geriatric Anxiety Inventory (GAS) aims to measure anxiety symptoms in the elderly in a dimensional way. The basic psychometric feature of the scale is that it can differentiate both the anxious/non-anxious group and the group with/without generalized anxiety disorder. The cut-off point of the scale for generalized anxiety disorder was determined as 10/11. Accordingly, the scale; "anxiety symptoms and generalized anxiety disorder > 10; only anxiety symptoms < 10". There is no reverse coded item in the scale, which consists of 20 items and is scored over two dimensions: "I agree" and "I do not agree". Accordingly, 1 point is given for the "agree" option and 0 points for the "disagree" option. Therefore, the scores obtained from the scale can vary between 0 and 20.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Assoc. Prof., Principal Investigator — Ordu Univercity
Locations (1):
- Hacer GOK UGUR, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cetin M, Gok Ugur H. The Effect of Flower Printing Activities on the Anxiety Levels of Elderly Nursing Home Residents: Randomized Controlled Study. Altern Ther Health Med. 2024 Oct;30(10):28-33. PMID 39316536